CLINICAL TRIAL: NCT03050827
Title: Muscarinic Receptor Antagonists as a Therapy for Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Aaron I. Vinik, MD, PhD, Director of Research & Neuroendocrine Unit, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-04-FB-0054
Record Dates: First submitted 2017-02-06; First posted 2017-02-13 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Diabetic; Neuropathic, Polyneuropathy (Manifestation)
MeSH Terms: conditions — Polyneuropathies | interventions — oxybutynin

STUDY DESIGN:
Intervention Model Description: The investigators propose a placebo controlled, double blinded study to examine efficacy of topical Gelnique 3%TM (3% oxybutynin) daily for 20 weeks) in improving IENF density in type 2 diabetic subjects with established peripheral neuropathy. Subjects with IENF loss of between 20-75% of normative values11 and thus amenable to therapy-induced recovery, will be randomized into placebo (N=30) or active drug (N=30) arms and instructed in how to apply 84 mg Gelnique 3%TM or hydrogel placebo to cover a 2 in2 region of skin adjacent to the initial biopsy site, as per the manufacturers instructions (http://www.gelnique.com/gel3/). Treatment will continue daily for 20 weeks, with monthly phone calls to monitor compliance. After 20 weeks, subjects will return for a second study visit and will undergo a series of measurements and 3 mm skin biopsy from the treated region of skin.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomizing and blinding an investigational drug will be done by assigning each patient/subject a study number in the order they are recruited. The patients are randomized using a randomizing web site at (www.randomizer.org). The randomized patient numbers are recorded. This code is then placed in an envelope and sealed. This envelope will remain sealed until the study is concluded. A blinding/randomization patient form will be completed for each patient and sealed in the individual envelopes. The outside of the envelopes will contain patient numbers for identification purposes. This will allow the research coordinator to break the individual blind in emergency situations without compromising the rest of the blinding data. All instances where the blind is broken will be documented appropriately.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3% oxybutynin (Active Comparator): Subjects with IENF loss of between 20-75% of normative values11 and thus amenable to therapy-induced recovery, will be randomized into the active drug arm (N=30) and instructed in how to apply 84 mg Gelnique 3%TM or hydrogel placebo to cover a 2 in2 region of skin adjacent to the initial biopsy site,
  Interventions: Drug: 3% oxybutynin
- Placebo (Placebo Comparator): Subjects with IENF loss of between 20-75% of normative values11 and thus amenable to therapy-induced recovery, will be randomized into the placebo group arm (N=30) and instructed in how to apply 84 mg Gelnique 3%TM or hydrogel placebo to cover a 2 in2 region of skin adjacent to the initial biopsy site,
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3% oxybutynin — Topical Gelnique 3%TM (3% oxybutynin) applied daily for 20 weeks in type 2 diabetic subjects with established peripheral neuropathy. Subjects will be randomized into placebo or active drug arms and instructed in how to apply 84 mg Gelnique 3%TM or hydrogel placebo to cover a 2 by 2 region of skin adjacent to the initial biopsy site. Treatment will continue daily for 20 weeks, with monthly phone calls to monitor compliance.
  Other Names: Gelnique 3%TM
  Arms: 3% oxybutynin
Drug: Placebo — Non-active placebo for 3% oxybutynin
  Arms: Placebo

SUMMARY:
Investigators propose a placebo controlled, double blinded study to examine efficacy of topical Gelnique 3%TM (3% oxybutynin) daily for 20 weeks) in improving IENF density in type 2 diabetic subjects with established peripheral neuropathy. This site most clearly demonstrated efficacy of topiramate in reversing IENF loss within 18 weeks in our prior study. Subjects will also undergo quantitative sensory testing (QST) and assays of laser Doppler skin blood flow (SkBF), neuropathy total symptom score (NTSS-6), and quality of life (Norfolk QOL-DN), along with standard measures of physiology and fasting blood chemistry. Subjects with IENF loss of between 20-75% of normative values and thus amenable to therapy-induced recovery, will be randomized into placebo (N=30) or active drug (N=30) arms and instructed in how to apply 84 mg Gelnique 3%TM or hydrogel placebo to cover a 2 in2 region of skin adjacent to the initial biopsy site, as per the manufacturers instructions (http://www.gelnique.com/gel3/). Treatment will continue daily for 20 weeks, with monthly phone calls to monitor compliance. After 20 weeks, subjects will return for a second series of measurements and 3 mm skin biopsy from the treated region of skin.

DETAILED DESCRIPTION:
Patient selection and characterization A total of 60 adults of both sexes and varying ethnicities, 30-80 years of age, will be recruited from Dr. Vinik's clinic. All participants will be diagnosed with established type 2 diabetes (>2 years) and diabetic peripheral neuropathy. Potential subjects will undergo a complete physical exam and a neurological exam to assess motor function and sensory perception28.

Randomizing and blinding an investigational drug will be done by assigning each patient/subject a study number in the order they are recruited. The patients are randomized using a randomizing web site at (www.randomizer.org). The randomized patient numbers are recorded. This code is then placed in an envelope and sealed. This envelope will remain sealed until the study is concluded. A blinding/randomization patient form will be completed for each patient and sealed in the individual envelopes. The outside of the envelopes will contain patient numbers for identification purposes. This will allow the research coordinator to break the individual blind in emergency situations without compromising the rest of the blinding data. All instances where the blind is broken will be documented appropriately.

Subject Recruitment Subjects of both sexes and all ethnicities will be recruited locally using the database of subjects available at The Strelitz Diabetes Research Center (SDRC) at Eastern Virginia Medical School (EVMS) as well as locally distributed flyers and notices, if needed. Approximately 60 randomized subjects are needed in this study to make a useful determination for current and future studies. Subjects who are dropped or withdraw from the study will be replaced.

Sample size estimation and data analysis:

Investigators have primarily powered the study based on variance data obtained in studies demonstrating efficacy of Topiramate on IENF density in diabetic subjects11. The sample size of 20 in each group (placebo vs. active drug) reflects the ability to detect a 20% deviation following treatment and was also sufficient to to identify therapy-induced improvements in SkBF and NTTS-6 score using a similar study design28. We intend to use ANOVA and MANOVA where data is normally distributed in raw form or in some cases after simple log-transformations. Based on these considerations, the 20 subjects in each group provide power greater than 0.80 for observing statistical significance at the p < 0.05 level. Relationships among measures of neurovascular function and changes in IENF will be determined with Spearman's rank correlation. If data are not normally distributed, the Wilcoxon signed-rank (within group) or Mann Whitney (between group) tests may be employed. The level of significance will be set at p<0.05.

FUTURE USE OF BIOLOGICAL SPECIMENS AND BANKING PROTOCOL After all of the required tests are finished, subjects will be asked if their leftover specimen may be stored for future research instead of throwing it away. Subjects will be asked to sign an addendum IRB approved consent form (#07-08-FB-0167) that allows the storage of biological specimen. An IRB application will be submitted for the use of any stored samples.

Study activity will take place after review and approval by the EVMS IRB (or other approved IRB). The IRB has the fundamental charge of protecting the rights and welfare of human participants in research. The EVMS Federal Wide Assurance assures that all research activities are guided by the ethical principles of The Belmont Report (respect for persons, beneficence, and justice) and activities comply with 45CFR46, regardless of funding source. These principles will be implemented through the process of informed consent by sharing information, ensuring subject comprehension and selecting volunteers without coercion or undue influence.

SAFETY EVALUATIONS AND ADVERSE EVENT REPORTING

Adverse events (AE's) will be recorded for all subjects. Relationship to study procedures performed will be documented by the investigator. Serious Adverse Events (SAEs) and pregnancies, which occur during this study, will be reported immediately upon their discovery to all appropriate agencies (Institutional Review Board (IRB). Serious Adverse Events are defined as any adverse event from this study that results in one of the following outcomes, or is significant for any other reason:

* Death
* Initial or prolonged inpatient hospitalization
* A life-threatening experience (that is, immediate risk of dying)
* Persistent or significant disability/incapacity
* Congenital anomaly/birth defect

The principal investigator will review the safety and progress of this study on a monthly basis. The principal investigator will review this protocol on a continuing basis for subject safety.

Risks and Protection Against Risk All subjects will be monitored for adverse and/or unexpected events. All information and data are kept in strict confidence. No information will be given to anyone without permission from the study participant.

Risks to participants will be minimized through subject selection, documented informed consent from the study participant, provisions made for the protection of privacy and confidentiality of data, and data monitoring to ensure subject safety. Data will be coded so that linkages to participants will only be available to the investigators. The database will be password protected and only the investigative staff will have access to the database. All subject names and personally identifiable data will be coded so that personal information (e.g., name, social security number, drivers' license number, address and phone number) remains private. Only the study investigators will have access to the information. Participants will not be personally identified in reports or publications.

Reproductive Risk Gelnique 3% is classified as a pregnancy category class B drug. Animal reproduction studies have failed to demonstrate a risk to the fetus and there are no adequate and well-controlled studies in pregnant women. Serum HcG testing for pregnancy will be performed at the screening. All participants will be asked to use birth control such as barrier methods (i.e. condoms, diaphragms), oral contraceptives, or intrauterine devices if they have not been surgically sterilized. Pregnancies will be treated as adverse events and will be followed to term.

Database Protection All data will be locally monitored according to the Strelitz Diabetes Center Standard Operating Procedures (see procedures below) and standard precautions will be made to protect personal health information.

1. Assign unique and secure User ID/password combination for each clinical research team member who has access to the computerized system(s). Ensure that users login using this unique User ID/password combination or other electronic signature when preparing to perform computer data entry or management functions.
2. Establish and maintain a schedule for changing each team member's User ID/password combination at appropriate intervals.
3. Invalidate stolen, lost or otherwise compromised User ID/password combinations and replace with a new combination.
4. Ensure that proper computer system function is routinely monitored.
5. Ensure that computerized systems are securely stored when not in use.
6. Log off when computer data entry/management activities are completed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of type 2 diabetes
* Participants between the ages of 30 and 80

Exclusion Criteria:

1. Presence of type 1 diabetes
2. Presence of renal insufficiency or pulmonary disease
3. Presence of clinically significant neuropathy that is clearly of non-diabetic origin
4. Amputations of lower extremities or presence of foot ulcers
5. Major macrovascular events such as myocardial infarction or stroke within the past 3 months
6. Uncontrolled or untreated hypothyroidism
7. Abnormalities of liver function defined as any liver enzymes (AST, ALT, SGPT, SGOT) greater than 3 times the upper limit of normal
8. Other serious medical conditions which, in the opinion of the investigator, would compromise the subject's participation in the study
9. Stable use (> 3 months) of antioxidant supplements or drugs known to affect oxidative stress and PDN
10. Allergy to oxybutynin or other ingredients in Gelnique 3%
11. Pregnancy or breastfeeding

13) History of alcohol abuse in the last year 14) Urinary retention or an enlarged prostate 15) Uncontrolled glaucoma 16) Gastric retention or gastroparesis (hard to digest food) 17) Currently taking other medicines to treat overactive bladder (Anticholinergics)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Intraepidermal Nerve Fiber Density | One Year
  Three mm skin biopsies will be taken at the two sites (lateral aspect of the proximal lower limb), on the non-dominant limb. Patients are pre-treated with 2% lidocaine with epinephrine and the biopsy is done with a sharp punch biopsy. All biopsy procedures are performed by a physician or physician's assistant under sterile conditions. Once removed the tissues are immediately transferred to storage buffer and frozen prior to sectioning and immunohistochemistry staining with PGP 9.5. Intraepidermal nerve fiber density and dendrite length. Sweat gland innervation in skin biopsies from diabetic subjects will also be determined. Sensitivity has been increased by using a 20 x 20 grid sampling system and our preliminary data shows correlation between IENF and sweat gland innervation in human skin biopsies.
Sudomotor Function | One Year
  Sudoscan will be used to measure the impact of reduced autonomic innervation of the sweat gland system using reverse iontophoresis. Sudoscan will employ sudorimetry to assess the sweat gland nerve fibers.
Ocular Nerve Fiber Density | One Year
  The investigators will use the Heidelberg Retina Tomograph (HRT) confocal corneal microscope. The corneal module will be used to study a very detailed view of cornea structure and pathology. Digital images of the patient's cornea will be taken with a microscope and laser scanning camera. A topical anesthetic (in the form of eye drops) will be used temporarily numb the cornea.

SECONDARY OUTCOMES:
Nerve Conduction Studies | One Year
  The XLtek Neuromax (XLtek, Inc., Ontario) and standard electrophysiological leads, stimulators, and techniques will be used for the nerve conduction tests. It is performed on the upper extremities (hands) and lower extremities (legs).
Quantitative Sensory Tests - Cold Pain Threshold | One Year
  The investigators will measure small fiber somatosensory function including cold pain thresholds at the dominant great toe, forearm, lateral aspect of proximal lower limb and finger in all subjects. Generally for each of these non-noxious sensations we will use the method of limits, 4 ascending trials with an inter-stimulus interval randomly varying from 4 to 20 seconds using the Medoc TSA 2001 / VSA 3000 (Medoc Advanced Medical, Minneapolis, MN).
Quantitative Sensory Tests - Heat Pain Threshold | One Year
  The investigators will measure small fiber somatosensory function including heat pain thresholds at the dominant great toe, forearm, lateral aspect of proximal lower limb and finger in all subjects. Generally for each of these non-noxious sensations we will use the method of limits, 4 ascending trials with an inter-stimulus interval randomly varying from 4 to 20 seconds using the Medoc TSA 2001 / VSA 3000 (Medoc Advanced Medical, Minneapolis, MN).
Quantitative Sensory Test - Cold Thermal Sensation | One Year
  The investigators will measure small fiber somatosensory function including cold thermal sensation at the dominant great toe, forearm, lateral aspect of proximal lower limb and finger in all subjects. Generally for each of these non-noxious sensations we will use the method of limits, 4 ascending trials with an inter-stimulus interval randomly varying from 4 to 20 seconds using the Medoc TSA 2001 / VSA 3000 (Medoc Advanced Medical, Minneapolis, MN).
Quantitative Sensory Tests - Warm Thermal Sensation | One Year
  The investigators will measure small fiber somatosensory function including warm thermal sensation at the dominant great toe, forearm, lateral aspect of proximal lower limb and finger in all subjects. Generally for each of these non-noxious sensations we will use the method of limits, 4 ascending trials with an inter-stimulus interval randomly varying from 4 to 20 seconds using the Medoc TSA 2001 / VSA 3000 (Medoc Advanced Medical, Minneapolis, MN).
Autonomic Function Tests - Standard Deviation of N-N interval | One Year
  The investigators will use the ANSAR device, which is the most sensitive measure of cardiac variation with respiration, to the standard deviation of N-N interval. This measurement will be used to separate sympathetic and parasympathetic function and relate these results to glabrous and hairy skin innervations.
Autonomic Function Tests - Root Mean Square of the Successive Differences | One Year
  The investigators will use the ANSAR device, which is the most sensitive measure of cardiac variation with respiration, to the Root Mean Square of the Successive Differences This measurement will be used to separate sympathetic and parasympathetic function and relate these results to glabrous and hairy skin innervations.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron I Vinik, MD, PhD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virgnia Medical School, Strelitz Diabetes Center, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Casselini CM, Parson HK, Frizzi KE, Marquez A, Smith DR, Guernsey L, Nemmani R, Tayarani A, Jolivalt CG, Weaver J, Fernyhough P, Vinik AI, Calcutt NA. A muscarinic receptor antagonist reverses multiple indices of diabetic peripheral neuropathy: preclinical and clinical studies using oxybutynin. Acta Neuropathol. 2024 Mar 25;147(1):60. doi: 10.1007/s00401-024-02710-4. PMID 38526612